CLINICAL TRIAL: NCT02983799
Title: Non-Randomized, Open-Label Phase II Study to Assess Olaparib Tablets as a Treatment for Subjects With Different HRD Tumor Status and With Platinum-Sensitive, Relapsed, High-Grade Serous or High-Grade Endometrioid Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer That Have Received at Least 1 Prior Line of Chemotherapy
Brief Title: Olaparib Tablets as a Treatment for Ovarian Cancer Subjects With Different HRD Tumor Status
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0816L00003
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2016-11-04; First posted 2016-12-06 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Relapsed Ovarian Cancer, BRCA Mutation, Platinum Sensitivity
Keywords: BRCA, ovarian, platinum, chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- gBRCAm; (Experimental): germline BRCA mutant
  Interventions: Drug: OLAPARIB
- sBRCAm and germline BRCA wild type; (Experimental): somatic BRCA mutant, germline BRCA wild type
  Interventions: Drug: OLAPARIB
- myChoice® HRD positive and BRCAwt; (Experimental): genomic instability positive and no BRCA mutation
  Interventions: Drug: OLAPARIB
- myChoice® HRD negative and BRCAwt (Experimental): genomic instability negative and no BRCA mutation
  Interventions: Drug: OLAPARIB

INTERVENTIONS:
Drug: OLAPARIB — 300 mg olaparib tablets taken orally twice daily

SUMMARY:
This is a non-randomized, open-label study to assess olaparib tablets as a treatment for subjects with different homologous recombination deficiency (HRD) tumor status and with platinum-sensitive, relapsed, high-grade serous or high-grade endometrioid ovarian cancer. Subjects should have received at least 1 prior line of platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is a Phase II, open-label, non-randomized, multi-center study assessing the efficacy and safety of olaparib tablets 300 mg (two 150 mg tablets) given orally twice daily (bid) in subjects with platinum-sensitive or partially platinum-sensitive, relapsed, high-grade serous or high-grade endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer, who have received at least 1 prior line of platinum-based chemotherapy.

The study will assess the effectiveness of olaparib tablets as measured by the objective response rate (ORR) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, in subjects with germline BRCA mutations (gBRCAm), somatic BRCA mutations (sBRCAm), or potential aberrations in homologous recombination deficiency (HRD) as determined by myChoice® HRD, as well as in subjects without identifiable HRD. This study will utilize Myriad BRACAnalysis CDx® for germline BRCA analysis and a tumor test (myChoice® HRD) for tumor BRCA analysis and HRD status. Four cohorts will be identified based upon the genetic testing described above:

* Cohort 1: gBRCAm,
* Cohort 2: sBRCAm and germline BRCA wild type,
* Cohort 3: myChoice® HRD positive (genomic instability positive) and BRCA wild type (BRCAwt) (no BRCA mutation),
* Cohort 4: myChoice® HRD negative (genomic instability negative) and BRCAwt (no BRCA mutation).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written signed informed consent prior to any study specific procedures;
* Female subjects with histologically diagnosed relapsed high-grade serous or high-grade endometrioid ovarian cancer;
* At least 1 lesion (measurable by RECIST v1.1) that can be accurately assessed at baseline by computed tomography (CT)/magnetic resonance imaging (MRI) and is suitable for repeated assessment;
* Subjects must have received at least 1 prior platinum-based line of chemotherapy for ovarian cancer. Note: There is no limit on the number of lines of chemotherapy;
* Subjects must be partially-platinum-sensitive (defined as progression 6 to 12 months after the end of the last platinum-based chemotherapy) or platinum sensitive (defined as progression > 12 months after the end of the last platinum-based chemotherapy);
* Subjects must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment;
* ECOG performance status 0 to 1;
* Subjects must have a life expectancy greater than or equal to 16 weeks;
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on Day 1;
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations; and
* Formalin fixed, paraffin embedded tumor sample (either archival or fresh sample) from the primary or recurrent cancer must be available for central testing. If there is not written confirmation of the availability of an archived or fresh tumor sample prior to enrollment, the subject is not eligible for the study.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca Representative staff and/or staff at the study site);
* Previous enrollment in the present study;
* Exposure to any investigational product (IP) within 30 days or 5 half-lives (whichever is longer) prior to start of study treatment;
* Any previous treatment with a PARP inhibitor, including olaparib;
* Subjects who have platinum-resistant or refractory disease defined as progression during or within 6 months of the last platinum-based chemotherapy;
* Other malignancy within the last 5 years (few exceptions apply);
* Resting ECG with clinically significant abnormal findings;
* Subjects receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment;
* Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors;
* Concomitant use of known strong or moderate CYP3A inducers;
* Persistent toxicities (> Common Terminology Criteria for Adverse Event [CTCAE] grade 2) caused by previous cancer therapy, excluding alopecia;
* Subjects with MDS/AML or with features suggestive of MDS/AML;
* Subjects with pneumonitis or at risk of pneumonitis;
* Subjects with symptomatic uncontrolled brain metastases;
* Major surgery within 2 weeks of starting study treatment, and subjects must have recovered from any effects of any major surgery;
* Subjects considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection;
* Breast feeding women;
* Immunocompromised subjects, e.g., subjects who are known to be serologically positive for human immunodeficiency virus;
* Subjects with known active hepatitis (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (32):
  - Research Site, Anchorage, Alaska
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, South Miami, Florida
  - Research Site, Skokie, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Silver Spring, Maryland
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Berkeley Heights, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Germantown, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Annandale, Virginia
  - Research Site, Milwaukee, Wisconsin
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Barnicle A, Ray-Coquard I, Rouleau E, Cadoo K, Simpkins F, Aghajanian C, Leary A, Poveda A, Lheureux S, Pujade-Lauraine E, You B, Ledermann J, Matulonis U, Gourley C, Timms KM, Lai Z, Hodgson DR, Elks CE, Dearden S, Egile C, Lao-Sirieix P, Harrington EA, Brown JS. Patterns of genomic instability in > 2000 patients with ovarian cancer across six clinical trials evaluating olaparib. Genome Med. 2024 Dec 18;16(1):145. doi: 10.1186/s13073-024-01413-5. PMID 39695768
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816L00003&attachmentIdentifier=1cc548a0-e0d8-4e45-a4e7-e90632b8c2cd&fileName=D0816L00003_SAP_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816L00003&attachmentIdentifier=4d8b8e75-6c5a-4aa7-aa28-8963de9d23cd&fileName=D0816L00003-CSP-V3__Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 272 subjects enrolled. One subject did not receive treatment and was excluded from analysis (Cohort 2 patient).
  All participants received a dose of 300mg BID of study drug
Groups:
- COHORT 1: germline BRCA mutant
- COHORT 2: somatic BRCA mutant, germline BRCA wild type
- COHORT 3: HRD positive and no BRCA mutation
- COHORT 4: HRD negative and no BRCA mutation
- Unassigned: Cohort unassigned
Period: Overall Study
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Unassigned
Started | 75 | 26 | 68 | 90 | 13
Completed (Patients continuing study at data cut-off) | 25 | 8 | 18 | 14 | 3
Not Completed | 50 | 18 | 50 | 76 | 10
Not completed — Withdrawn from study before data cut-off | 28 | 12 | 23 | 25 | 1
Not completed — Death | 20 | 5 | 23 | 47 | 7
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 4 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Unassigned | Total
Number analyzed (Participants) | 75 | 26 | 68 | 90 | 13 | 272
Age, Continuous [Mean (Standard Deviation); unit: Age Continuous] — Population: A total of 272 subjects enrolled. One subject did not receive treatment and was excluded from analysis (Cohort 2 patient).
  Age Continuous
    number analyzed (Participants) | 75 | 25 | 68 | 90 | 13 | 271
    (all) | 60.7 (9.3) | 69.7 (9.0) | 63.2 (9.9) | 67.8 (9.5) | 69.8 (10.0) | 64.9 (10.1)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 75 | 26 | 68 | 90 | 13 | 272
Race/Ethnicity, Customized [Number; unit: Participants]
  WHITE | 58 | 23 | 50 | 78 | 11 | 220
  BLACK OR AFRICAN AMERICAN | 7 | 0 | 5 | 5 | 0 | 17
  ASIAN | 6 | 3 | 11 | 6 | 2 | 28
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0 | 0 | 0 | 0
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 1 | 0 | 0 | 1
  OTHER | 4 | 0 | 1 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate, Defined as the Percentage of Subjects With a Best Overall Response of Confirmed Complete Response (CR) or Partial Response (PR)
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using ORR according to RECIST v1.1 criteria (Investigator determined)
Time Frame: From first dose up until progression, or last evaluable assessment in the absence of progression (up to 36 months)
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Cohort 1 | Cohort 2 | COHORT 3 | COHORT 4 | Unassigned
Number analyzed (Participants) | 75 | 25 | 68 | 89 | 13
Percent | 69.3 [57.6 to 79.5] | 64.0 [42.5 to 82.0] | 29.4 [19.0 to 41.7] | 10.1 [4.7 to 18.3] | 30.8 [9.1 to 61.4]

2. Secondary Outcome: Duration of Response, for Those Subjects With a Confirmed Response of CR or PR
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using duration of response
Time Frame: From the date of the measurement criteria for CR or PR are first met until the date of documented progression or death in the absence of disease progression (up to 36 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | COHORT 3 | COHORT 4 | Unassigned
Number analyzed (Participants) | 52 | 16 | 20 | 9 | 4
Months | 9.4 [7.5 to 12.5] | 14.7 [5.7 to NA] — Not estimable due to limited data. | 10.0 [5.6 to NA] — Not estimable due to limited data. | 5.3 [3.7 to 7.3] | 7.5 [6.0 to NA] — Not estimable due to limited data.

3. Secondary Outcome: CA-125 Response Rate, Defined as the Percentage of Subjects With a CA-125 Response According to GCIG Criteria Divided by the Number of Subjects Evaluable for CA-125 Response
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using CA-125 response rate
Time Frame: From baseline to Day 1 of each cycle and end of study treatment visit (up to 36 months)
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Cohort 1 | Cohort 2 | COHORT 3 | COHORT 4 | Unassigned
Number analyzed (Participants) | 44 | 20 | 48 | 64 | 12
Percent | 93.2 [81.3 to 98.6] | 70.0 [45.7 to 88.1] | 47.9 [33.3 to 62.8] | 26.6 [16.3 to 39.1] | 66.7 [34.9 to 90.1]

4. Secondary Outcome: Disease Control Rate Defined as the Percentage of Subjects Who Have a Best Overall Response of CR or PR or SD at Greater Than or Equal to 8 Weeks Divided by the Number of Subjects in the Efficacy Analysis Set, Prior to Any PD Event
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using disease control rate (DCR). DCR is defined as the percentage of subjects with a best overall response of CR or PR (at any time up to and including the defined analysis cut-off point) or who have demonstrated stable disease (SD) for at least 8 weeks from first dose, divided by the number of subjects in the efficacy analysis set.
Time Frame: From first dose up until progression, or last evaluable assessment in the absence of progression
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Cohort 1 | Cohort 2 | COHORT 3 | COHORT 4 | Unassigned
Number analyzed (Participants) | 75 | 25 | 68 | 89 | 13
Percent | 96.0 [88.8 to 99.2] | 100.0 [86.3 to 100.0] | 79.4 [67.9 to 88.3] | 75.3 [65.0 to 83.8] | 92.3 [64.0 to 99.8]

5. Secondary Outcome: Progression Free Survival
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using progression free survival
Time Frame: From first dose to earlier date of assessment of objective progression or death by any cause in the absence of progression (up to 36 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | COHORT 3 | COHORT 4 | Unassigned
Number analyzed (Participants) | 75 | 25 | 68 | 89 | 13
Months | 11 [8.3 to 12.2] | 10.8 [7.3 to NA] — Not estimable due to limited data. | 7.2 [5.3 to 7.6] | 5.4 [3.7 to 5.6] | 9.2 [3.5 to 12.7]

6. Secondary Outcome: Time to Any Progression
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using time to any progression
Time Frame: From first dose to earlier date of CA-125 progression or RECIST v1.1 progression, or death by any cause in absence of progression (up to 36 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | COHORT 3 | COHORT 4 | Unassigned
Number analyzed (Participants) | 75 | 25 | 68 | 89 | 13
Months | 10.9 [7.4 to 13.3] | 11.1 [6.6 to NA] — Not estimable due to limited data. | 7.2 [3.8 to 7.6] | 5.3 [3.7 to 5.5] | 7.3 [3.5 to 9.7]

7. Secondary Outcome: Overall Survival
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using overall survival
Time Frame: From date of first dose to date of death from any cause (up to 48 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | COHORT 3 | COHORT 4 | Unassigned
Number analyzed (Participants) | 75 | 25 | 68 | 89 | 13
Months | NA [29.2 to NA] — Not estimable due to limited data. | NA [NA to NA] — Not estimable due to limited data. | NA [22.8 to NA] — Not estimable due to limited data. | 23.8 [16.6 to 31.4] | 18 [8 to NA] — Not estimable due to limited data.

8. Secondary Outcome: HRD Status as Per HRRm Gene Panel Assessment Will be Correlated With Clinical Outcome (ORR) for Subjects Enrolled in the 2 Cohorts With BRCAwt (Cohorts 3 and 4)
Description: To determine the clinical effectiveness of olaparib treatment in each of 4 cohorts assessed using HRRm gene panel status related to clinical outcome
Time Frame: At baseline
Measure: Number (95% Confidence Interval); unit: Percent
Groups:
- Cohort 3, HRRm Pos: HRD positive and no BRCA mutation, HRRm positive
- Cohort 3, HRRm Neg: HRD positive and no BRCA mutation, HRRm negative
- Cohort 4, HRRm Pos: HRD negative and no BRCA mutation, HRRm positive
- Cohort 4, HRRm Neg: HRD negative and no BRCA mutation, HRRm negative
Arm/Group | Cohort 3, HRRm Pos | Cohort 3, HRRm Neg | Cohort 4, HRRm Pos | Cohort 4, HRRm Neg
Number analyzed (Participants) | 9 | 56 | 12 | 76
Percent | 11.1 [0.3 to 48.2] | 32.1 [20.3 to 46.0] | 8.3 [0.2 to 38.5] | 10.5 [4.7 to 19.7]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs), serious AEs, AEs of special interest (AESIs), and AEs leading to discontinuation were collected from signature of informed consent for study participation. Treatment emerging AEs were reported from date of first dose of study treatment and continued throughout the active treatment period and the follow-up period 30 days after the last dose of olaparib. After the primary analysis data cut-off till study completion, only deaths, SAEs, AESIs and DAEs were collected/reported.
Description: Adverse events and serious adverse events are reported in the safety analysis set including all patients who received at least one dose of study treatment. Between the primary analysis data cut-off and final data cut-off (12-month overall survival), only serious adverse events, adverse events of special interest, and adverse events leading to discontinuation were collected.
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | UNASSIGNED
All-Cause Mortality (participants affected / at risk) | 20/75 | 5/25 | 23/68 | 47/90 | 7/13
Serious Adverse Events (participants affected / at risk) | 13/75 | 8/25 | 7/68 | 35/90 | 6/13
Other Adverse Events (participants affected / at risk) | 75/75 | 25/25 | 67/68 | 88/90 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=75) | COHORT 2 (N=25) | COHORT 3 (N=68) | COHORT 4 (N=90) | UNASSIGNED (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 6 (7) | 4 (6)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Strangulated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hydroureter (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=75) | COHORT 2 (N=25) | COHORT 3 (N=68) | COHORT 4 (N=90) | UNASSIGNED (N=13)
Anaemia (Blood and lymphatic system disorders) | 18 (25) | 7 (13) | 14 (16) | 31 (38) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0) | 2 (3) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 11 (12) | 2 (4) | 9 (10) | 8 (8) | 1 (3)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 15 (20) | 4 (4) | 10 (10) | 13 (17) | 7 (9)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 6 (8) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (8) | 1 (2)
Breath odour (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (19) | 7 (8) | 19 (19) | 24 (28) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 17 (23) | 4 (4) | 15 (20) | 18 (25) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 8 (8) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 3 (4) | 9 (10) | 11 (11) | 4 (5)
Eructation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (6) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (18) | 2 (2) | 5 (6) | 7 (8) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 50 (84) | 20 (38) | 42 (66) | 60 (76) | 8 (11)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 21 (37) | 12 (17) | 15 (27) | 35 (56) | 6 (10)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (6) | 0 (0)
Early satiety (General disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 50 (55) | 15 (16) | 43 (46) | 50 (56) | 9 (13)
Feeling cold (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 3 (4) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 10 (11) | 4 (4) | 3 (3) | 14 (24) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 1 (1)
Suprapubic pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Laryngitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (12) | 1 (2) | 3 (3) | 6 (6) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Oral herpes (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin candida (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (15) | 3 (4) | 5 (5) | 11 (12) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (6) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3) | 2 (3) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 10 (10) | 9 (18) | 13 (14) | 13 (16) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Carbohydrate antigen 125 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 4 (5) | 2 (2) | 4 (4) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 0 (0) | 4 (5) | 1 (1) | 1 (2)
Platelet count decreased (Investigations) | 3 (5) | 1 (1) | 3 (5) | 2 (2) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 4 (4) | 6 (8) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (4) | 0 (0) | 2 (5) | 2 (2) | 1 (2)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (14) | 6 (6) | 16 (16) | 21 (25) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (8) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 4 (6) | 4 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 5 (5) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 2 (2) | 5 (6) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (2) | 5 (5) | 8 (9) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 4 (6) | 4 (4) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4) | 4 (5) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 3 (3) | 7 (8) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 10 (10) | 7 (10) | 11 (14) | 12 (14) | 1 (2)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 7 (7) | 5 (5) | 13 (15) | 14 (14) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 2 (3) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 3 (4) | 0 (0) | 2 (2) | 3 (4) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (1) | 6 (7) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 5 (5) | 1 (1) | 2 (2) | 4 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vaginal lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (4) | 12 (14) | 14 (14) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 4 (5) | 8 (9) | 20 (22) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 2 (2) | 5 (5) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Collateral circulation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 0 (0) | 8 (8) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2) | 2 (2) | 3 (4) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 19 (28) | 8 (10) | 13 (17) | 11 (13) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and PI shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within two (2) years of completion of the Study shall require the Sponsor's prior written consent. Sponsor to be consulted prior to presentation or publication.

DOCUMENTS (2):
  • Study Protocol (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT02983799/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT02983799/SAP_001.pdf